CLINICAL TRIAL: NCT05845151
Title: Fibroblast Activating Protein Inhibitor PET Imaging for Molecular Assessment of Fibroblast Activation and Risk Evaluation in Patients With Lupus Nephritis
Brief Title: Fibroblast Activating Protein Inhibitor PET Imaging in Lupus Nephritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: (2021)CER(87)
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LN Patients group (Experimental)
  Interventions: Diagnostic Test: 68Ga-FAPI-04 PET

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-04 PET — Activation of renal fibroblast is quantified using 68Ga-FAPI-04 PET in patients with LN.

SUMMARY:
Abnormal high expression of fibroblast activating protein (FAP) has been found in inflammatory reactions and benign fibrosis tissue. Autoimmune nephropathy such as lupus nephritis (LN) can lead to tubular atrophy and excessive deposition of extracellular matrix, which may be accompanied by abnormally increased expression of activated FAP in kidney tissue, and lead to renal fibrosis and long-term renal failure. This makes 68Ga-labeled FAP inhibitor (FAPI) positron emission tomography (PET) imaging the potential to early assess disease severity, predict disease progress and aid treatment planning in patients with LN. Compared to renal pathological puncture, 68Ga-FAPI PET is a new tool for non-invasive, repeatable assessment of renal fibrotic activation.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18-80 years old;
* Confirmed SLE: meet the 2019 EULAR/ACR classification standards;
* There are signs of renal involvement and indications for renal puncture: proteinuria> 0.5g/24 hours (or urine protein creatine ratio (UPCR) >500mg/g), unexplained decrease of glomerular filtration rate (GFR)

Exclusion Criteria:

* The pathology of renal puncture is not consistent with lupus nephritis;
* Previous history of other kidney diseases;
* There are contraindications to renal puncture: (1) obvious bleeding tendency, (2) severe hypertension, (3) psychosis or non-cooperative patients, (4) isolated kidney, (5) small kidney;
* History of malignant tumors within 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Renal FAP expression level | Baseline
  Quantitative assessment of renal fibroblast activation on FAPI PET image
Renal FAP expression level | 6 months after baseline
  Quantitative assessment of renal fibroblast activation on FAPI PET image
Renal FAP expression level | 12 months after baseline
  Quantitative assessment of renal fibroblast activation on FAPI PET image
Renal FAP expression level | 24 months after baseline
  Quantitative assessment of renal fibroblast activation on FAPI PET image

SECONDARY OUTCOMES:
Renal fibrosis score | Baseline
  It's an immunohistochemical staining-based score after renal puncture. Higher score means a worse outcome.
Chronic activity score | Baseline
  It's an immunohistochemical staining-based scores after renal puncture. Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Shi, Dr., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, China